CLINICAL TRIAL: NCT00618072
Title: EMPOWIR: Enhance the Metabolic Profile of Women With Insulin Resistance: Carbohydrate Modified Diet Alone and in Combination With Metformin or Metformin Plus Avandia in Non-diabetic Women With Midlife Weight Gain and Documented Insulin Elevations (Syndrome W)
Brief Title: EMPOWIR:Enhance the Metabolic Profile of Women With Insulin Resistance
Acronym: EMPOWIR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: New York Medical College (Other)
Collaborators: Albert Einstein College of Medicine (Other); University of Tennessee (Other)
Responsible Party: Principal Investigator, Harriette Mogul, Director Research< Division of Adult Endocrinology, New York Medical College
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GSK-109157; GSK CRN: 007674
Record Dates: First submitted 2008-02-05; First posted 2008-02-18 (Estimated); Results first posted 2014-03-28 (Estimated); Last update posted 2014-03-28 (Estimated); Status verified 2014-03

CONDITIONS: Hyperinsulinemia; Insulin Resistance; Obesity
Keywords: hyperinsulinemia; insulin resistance; perimenopause; obesity; overweight; women
MeSH Terms: conditions — Hyperinsulinism; Insulin Resistance; Obesity; Overweight | interventions — rosiglitazone-metformin combination; Metformin; Rosiglitazone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A: Study diet (Placebo Comparator): EMPOWIR dietary intervention food exchange program; 40-45% carbohydrates, 35-40% protein, and 20% fat AND 4 week dosage escalation of placebo metformin, 500 mg/day to a total dose of 2000mg/day; starting dose of placebo rosiglitazone 2mg/day added at weeks 3 and weeks 4 to a total dose of 4 mg/day.
  Interventions: Drug: metformin and rosiglitazone
- B: Study diet plus Metformin (Active Comparator): Metformin and Rosiglitazone Placebo
  EMPOWIR dietary intervention food exchange program; 40-45% carbohydrates, 35-40% protein, and 20% fat AND 4 week dosage escalation of metformin, 500 mg/day to a total dose of 2000mg/day; starting dose of placebo rosiglitazone 2mg/day added at weeks 3 and weeks 4 to a total dose of 4 mg/day.
  Interventions: Drug: metformin and rosiglitazone
- C: Study diet plus metformin and avandia (Active Comparator): Metformin and Rosiglitazone
  EMPOWIR dietary intervention food exchange program; 40-45% carbohydrates, 35-40% protein, and 20% fat AND 4 week dosage escalation of metformin, 500 mg/day to a total dose of 2000mg/day; starting dose of rosiglitazone 2mg/day added at weeks 3 and weeks 4 to a total dose of 4 mg/day.
  Interventions: Drug: metformin and rosiglitazone

INTERVENTIONS:
Drug: metformin and rosiglitazone — 4 week dosage escalation of metformin, 500 mg/day (or placebo) to a total dose of 2000mg/day; starting dose of rosiglitazone 2mg/day(or placebo) added at weeks 3 and weeks 4 to a a total dose of 4 mg/day
  Other Names: glucophage; avandia; avandamet

SUMMARY:
The goal of the study is to identify and treat women with midlife weight gain who have normal blood sugars, but increased insulin levels (hyperinsulinemia) following the performance of a glucose tolerance test. The study will evaluate effects of a unique carbohydrate modified diet alone and in combination with metformin(MF) and Avandamet® (MF plus rosiglitazone (RSG)) on insulin levels in a wide range of ethnically diverse women (aged 35-55) at three academic medical centers. The primary study hypothesis is that insulin sensitizing medications, in combination with alterations in carbohydrate intake, will reduce insulin levels and improve established risk factors for the metabolic syndrome.

The alarming prevalence of obesity, diabetes, and related comorbidities and the paucity of easily adopted, cost-effective preventive strategies for high risk populations, suggest that pharmaco-therapies and dietary regimens targeted to reducing insulin resistance could have important clinical and public health implications.

DETAILED DESCRIPTION:
Progressive weight gain that starts in the fourth and fifth decades is commonly reported by women from all ethnic and socio-economic groups. Our previous data suggest that, in large and diverse subpopulations of healthy-appearing women this midlife weight gain may represent the earliest clinical manifestation of insulin resistance - demarcated by increased insulin response curves in the presence of completely normal glucose tolerance tests. We termed the disorder Syndrome W to highlight its defining triad of weight gain, waist gain and white-coat hypertension in women and its role as an alphabetic and chronologic antecedent to the better known Syndrome X. As in other disorders of insulin action in younger women, including Polycystic Ovarian Syndrome (PCOS), early adrenarche, and precocious puberty, Syndrome W is, presumably, a harbinger of The Metabolic Syndrome and Type 2 diabetes at an early and optimal period for intervention.

Preliminary data from our first pilot study suggested that metformin, in combination with a hypocaloric, low-fat, carbohydrate modified dietary program produced significant and sustainable weight loss in women with Syndrome W, with notable reductions in fasting insulin levels. These findings supported hypotheses that insulin elevation might be an antecedent, as well as a consequence, of weight gain, accounting for a progressive and intractable weight spiral as women transition from their forties to their sixties. Additional two to four year follow-up in an intention-to-treat analysis of consecutive women who lost ≥10% of their body weight after one year of the treatment regimen further suggests that this composite intervention prevents weight regain and the onset of overt glucose impairment. The protocol evolved from evaluation and treatment of several hundred patients seen in The Endocrine Faculty Practice over a ten year period and has been highly successful in a broad ethnic range of normo-glycemic, hyperinsulinemic subjects. These include midlife women with weight gain and overweight men with upper body obesity - populations which have not been comparably treated in prior studies which focus predominantly on subjects with discernible glycemic abnormalities. The magnitude and duration of the treatment effect suggest that more rigorous study should be undertaken with a randomized clinical trial.

PPAR agonists including thiazolidinediones (TZD's) are a newer category of insulin sensitizers with increasingly wide and well-studied positive attributes, including redistribution of fat depots, increased adiponectin secretion, and reduction of inflammatory and proinflammatory markers.

The combination of metformin and rosiglitazone (Avandamet®) is FDA-approved for the treatment of hyperglycemia in patients with Type 2 diabetes. Previous clinical research and recent laboratory data suggest that the two categories of insulin sensitizers have independent and additive mechanisms of action that could target and, ultimately, modulate the underlying pathogenesis of insulin resistance.

Comparison studies suggest that TZD's may have a greater insulin sensitizing action and provide greater reduction in hyperinsulinemia than metformin. However, due to increased adipocyte expression (and possible other mechanisms), weight gain is a common and undesirable side effect of TZD treatment. The addition of metformin to rosiglitazone, along with dietary strategies that reduce endogenous insulin production could prove an ideal therapeutic option to attenuate insulin resistance and preserve ß-cell function in high risk individuals. Early initiation of this dual regimen in normoglycemic subjects with documented hyperinsulinemia could have profound implications for Syndrome W women and for an additional 25% of the adult US population estimated to have other manifestations of The Metabolic Syndrome.

The primary study question addressed is whether dual treatment regimens which modulate insulin action can reduce hyperinsulinemia and insulin resistance in high risk, but healthy-appearing normoglycemic, hyperinsulinemic subjects identified because of progressive, intractable, midlife weight gain

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, non-diabetic women with "≥20 pound weight gain since their twenties"
2. Age: 35-55
3. Peri-menopausal or postmenopausal status
4. Body Mass Index (BMI) 25-35 kg/m2
5. Either:

   1. a single blood pressure recording ≥135/85 or the use of blood pressure medication OR
   2. HDL≤50mg/dl or triglycerides ≥150 mg/dl or the use of lipid modifying medication
6. Area-under-the-curve (AUC-)insulin level>100mcgU/ml along with normal fasting (≤100 mg/dl) & postprandial ((≤200 mg/dl) glucose determinations following a 75-gram standard oral glucose tolerance test.

   -

Exclusion Criteria:

1. known diabetes, fasting blood sugar ≥100 mg/dl or HbA-1-C≥6.0%
2. known hepatic disease or ALT>40
3. known renal disease or creatinine ≥ 1.4
4. known severe pulmonary disease
5. chronic acidosis of any etiology
6. Congestive heart failure (NYS Category 1), treated or untreated
7. Cancer - active within 5 years
8. current alcoholism or other substance abuse
9. co-morbid psychiatric disorder, which in the opinion of the screening physician would require concomitant psychotherapy as part of obesity management
10. currently untreated thyroid abnormality (TSH≤0.2 or ≥4mIU/L)
11. pregnancy or contemplation of pregnancy
12. use of TZD or metformin within the past year
13. allergy to TZD or biguanide
14. use of FDA approved or alternate obesity agent within 6 months of the study
15. history of pseudotumor cerebri
16. other impairment, such as a history of medication noncompliance, which in the judgment of the screening clinician, would preclude active study participation.
17. history of known or suspected heart disease

Ages: 35 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2008-01; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harriette R Mogul, MD MPH, Principal Investigator — New York Medical College
Locations (1):
- Albert Einstein College of Medicine, The Bronx, New York, United States

REFERENCES:
- [Background] Mogul HR, Peterson SJ, Weinstein BI, Zhang S, Southren AL. Metformin and carbohydrate-modified diet: a novel obesity treatment protocol: preliminary findings from a case series of nondiabetic women with midlife weight gain and hyperinsulinemia. Heart Dis. 2001 Sep-Oct;3(5):285-92. doi: 10.1097/00132580-200109000-00002. PMID 11975807
- [Background] Mogul HR, Weinstein BI, Mogul DB, Peterson SJ, Zhang S, Frey M, Gambert SR, Southren AL. Syndrome W: a new model of hyperinsulinemia, hypertension and midlife weight gain in healthy women with normal glucose tolerance. Heart Dis. 2002 Mar-Apr;4(2):78-85. doi: 10.1097/00132580-200203000-00004. PMID 11975838
- [Background] Mogul HR, Peterson SJ, Weinstein BI, Li J, Southren AL. Long-term (2-4 year) weight reduction with metformin plus carbohydrate-modified diet in euglycemic, hyperinsulinemic, midlife women (Syndrome W). Heart Dis. 2003 Nov-Dec;5(6):384-92. doi: 10.1097/01.hdx.0000098361.84908.9c. PMID 14633321
- [Background] Mogul HR, Marshall M, Frey M, Burke HB, Wynn PS, Wilker S, Southern AL, Gambert SR. Insulin like growth factor-binding protein-1 as a marker for hyperinsulinemia in obese menopausal women. J Clin Endocrinol Metab. 1996 Dec;81(12):4492-5. doi: 10.1210/jcem.81.12.8954066.
- [Derived] Mogul H, Freeman R, Nguyen K. METFORMIN-SUSTAINED WEIGHT LOSS AND REDUCED ANDROID FAT TISSUE AT 12 MONTHS IN EMPOWIR (ENHANCE THE METABOLIC PROFILE OF WOMEN WITH INSULIN RESISTANCE): A DOUBLE BLIND, PLACEBO-CONTROLLED, RANDOMIZED TRIAL OF NORMOGLYCEMIC WOMEN WITH MIDLIFE WEIGHT GAIN. Endocr Pract. 2016 May;22(5):575-86. doi: 10.4158/EP151087.OR. Epub 2016 Jan 20. PMID 26789348
- [Derived] Mogul HR, Freeman R, Nguyen K, Frey M, Klein LA, Jozak S, Tanenbaum K. Carbohydrate modified diet & insulin sensitizers reduce body weight & modulate metabolic syndrome measures in EMPOWIR (enhance the metabolic profile of women with insulin resistance): a randomized trial of normoglycemic women with midlife weight gain. PLoS One. 2014 Sep 26;9(9):e108264. doi: 10.1371/journal.pone.0108264. eCollection 2014. PMID 25259787

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled from December 2007 until November 2010. The study was conducted at two academic medical centers: Montefiore Hospital/Einstein, Bronx, and Westchester Medical Center/New York Medical College, Valhalla, NY in conjunction with the GCRC at Einstein.
Pre-assignment Details: Prior to randomization, subjects attended 4 weekly workshops to introduce study instruments & the EMPOWIR diet -a food exchange program promoting intake of vegetables, low-glycemic index fruits, low-fat protein & dairy products, elimination of added sugars & the notable restriction of 3 additional allowable carbohydrates to after 4PM.
Groups:
- A: EMPOWIR Diet and Placebo: EMPOWIR dietary intervention food exchange program; 40-45% carbohydrates, 35-40% protein, and 20% fat AND 4 week dosage escalation of placebo metformin, 500 mg/day to a total dose of 2000mg/day; starting dose of placebo rosiglitazone 2mg/day added at weeks 3 and weeks 4 to a total dose of 4 mg/day.
- B: EMPOWIR Diet Plus Metformin and Placebo Avandia; C: EMPOWIR Diet Plus Metformin and Avandia: EMPOWIR dietary intervention food exchange program; 40-45% carbohydrates, 35-40% protein, and 20% fat AND 4 week dosage escalation of metformin, 500 mg/day to a total dose of 2000mg/day; starting dose of placebo rosiglitazone 2mg/day added at weeks 3 and weeks 4 to a total dose of 4 mg/day.
Period: Overall Study
Arm/Group | A: EMPOWIR Diet and Placebo | B: EMPOWIR Diet Plus Metformin and Placebo Avandia | C: EMPOWIR Diet Plus Metformin and Avandia
Started | 16 | 15 | 15
Completed | 14 | 14 | 11
Not Completed | 2 | 1 | 4
Not completed — Lost to Follow-up | 2 | 0 | 3
Not completed — Physician Decision | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- C: EMPOWIR Diet Plus Metformin and Avandia: EMPOWIR dietary intervention food exchange program; 40-45% carbohydrates, 35-40% protein, and 20% fat AND 4 week dosage escalation of metformin, 500 mg/day to a total dose of 2000mg/day; starting dose of rosiglitazone 2mg/day added at weeks 3 and weeks 4 to a total dose of 4 mg/day
- Total: Total of all reporting groups
Arm/Group | A: EMPOWIR Diet and Placebo | B: EMPOWIR Diet Plus Metformin and Placebo Avandia | C: EMPOWIR Diet Plus Metformin and Avandia | Total
Number analyzed (Participants) | 16 | 15 | 15 | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 16 | 15 | 15 | 46
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 15 | 15 | 46
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 16 | 15 | 15 | 46
Fasting insulin [Mean (Standard Deviation); unit: uIU/mL] | 11.2 (1.4) | 12.5 (2.0) | 8.7 (1.5) | 10.7 (0.7)
Body Weight [Mean (Standard Deviation); unit: kg] | 84.1 (2.8) | 85.1 (2.4) | 81.8 (3.2) | 82.4 (1.63)
HOMA-IR [Mean (Standard Deviation); unit: HOMA-IR score] | 2.3 (0.2) | 2.5 (0.4) | 1.9 (0.3) | 2.3 (0.2)
Waist circumference [Mean (Standard Deviation); unit: cm] | 97.5 (2.3) | 92.9 (1.8) | 93.1 (2.1) | 94.7 (1.27)
Systolic BP [Mean (Standard Deviation); unit: mmHg] | 117.5 (2.9) | 114.3 (3.4) | 118.7 (6.0) | 118.2 (2.1)
Diastolic BP [Mean (Standard Deviation); unit: mmHg] | 75.9 (2.6) | 75.3 (2.0) | 76.9 (4.2) | 75.4 (1.4)
HDL [Mean (Standard Deviation); unit: mg/dl] | 49.3 (2.3) | 61.6 (5.7) | 60.1 (3.2) | 58.9 (2.4)
Triglycerides [Mean (Standard Deviation); unit: mg/dl] | 90.1 (9.5) | 88.0 (11.3) | 82.6 (11.2) | 86.9 (9.3)
Adiponectin [Mean (Standard Deviation); unit: ug/mL] | 9.3 (1.3) | 10.6 (1.4) | 11.1 (1.0) | 10.6 (4.6)

OUTCOME MEASURES:

1. Primary Outcome: Fasting Insulin
Description: Insulin was determined with a Siemens Immulite assay with respective intra-and inter-CV's 5.7 and 5.9%, and no cross reactivity to pro-insulin.
Time Frame: 6 months
Population: The final data-set consisted of 44 study participants, after exclusion of two study completers due to clinical conditions which appeared de novo (asthma requiring high dose prednisone and growth hormone deficiency diagnosed mid-study) - applicable to all study outcomes.
Measure: Mean (Standard Error); unit: uIU/mL
Arm/Group | A: EMPOWIR Diet and Placebo | B: EMPOWIR Diet Plus Metformin and Placebo Avandia | C: EMPOWIR Diet Plus Metformin and Avandia
Number analyzed (Participants) | 16 | 14 | 14
uIU/mL | 8.1 (1.3) | 8.0 (1.2) | 6.3 (0.9)
Statistical Analysis 1: Comparison: A: EMPOWIR Diet and Placebo; Paired t-tests were used to compare within-group mean differences at baseline and at 6 months following randomization for each of the 3 comparator groups; Test type: Superiority or Other; p = 0.181, Paired t-test
Statistical Analysis 2: Comparison: B: EMPOWIR Diet Plus Metformin and Placebo Avandia; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.026, Paired t-test
Statistical Analysis 3: Comparison: C: EMPOWIR Diet Plus Metformin and Avandia; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.063, Paired t-test

2. Secondary Outcome: Body Weight
Description: Body weight measurement was performed three times and averaged by a single study coordinator.
Time Frame: 6 months
Measure: Mean (Standard Error); unit: kg
Arm/Group | A: EMPOWIR Diet and Placebo | B: EMPOWIR Diet Plus Metformin and Placebo Avandia | C: EMPOWIR Diet Plus Metformin and Avandia
Number analyzed (Participants) | 16 | 14 | 14
kg | 80.0 (2.7) | 80.4 (2.1) | 77.5 (4.0)
Statistical Analysis 1: Comparison: A: EMPOWIR Diet and Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.049, Paired t-test
Statistical Analysis 2: Comparison: B: EMPOWIR Diet Plus Metformin and Placebo Avandia; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.002, Paired t-test
Statistical Analysis 3: Comparison: C: EMPOWIR Diet Plus Metformin and Avandia; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.032, Paired t-test

3. Secondary Outcome: HOMA-IR
Description: HOMA-IR was calculated by the formula: fasting insulin (uU/mL) times fasting glucose (mg/L) divided by 22.5.
Time Frame: 6 months
Measure: Mean (Standard Error); unit: HOMA-IR score
Arm/Group | A: EMPOWIR Diet and Placebo | B: EMPOWIR Diet Plus Metformin and Placebo Avandia | C: EMPOWIR Diet Plus Metformin and Avandia
Number analyzed (Participants) | 16 | 14 | 14
HOMA-IR score | 1.5 (0.1) | 1.6 (0.3) | 1.3 (0.2)
Statistical Analysis 1: Comparison: A: EMPOWIR Diet and Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.142, Paired t-test
Statistical Analysis 2: Comparison: B: EMPOWIR Diet Plus Metformin and Placebo Avandia; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.054, Paired t-test
Statistical Analysis 3: Comparison: C: EMPOWIR Diet Plus Metformin and Avandia; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.013, Paired t-test

4. Secondary Outcome: Waist Circumference
Time Frame: 6 months
Measure: Mean (Standard Error); unit: cm
Arm/Group | A: EMPOWIR Diet and Placebo | B: EMPOWIR Diet Plus Metformin and Placebo Avandia | C: EMPOWIR Diet Plus Metformin and Avandia
Number analyzed (Participants) | 16 | 14 | 14
cm | 93.1 (2.1) | 90.4 (1.9) | 87.5 (3.2)
Statistical Analysis 1: Comparison: A: EMPOWIR Diet and Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.052, Paired t-test
Statistical Analysis 2: Comparison: B: EMPOWIR Diet Plus Metformin and Placebo Avandia; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.143, Paired t-test
Statistical Analysis 3: Comparison: C: EMPOWIR Diet Plus Metformin and Avandia; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.005, Paired t-test

5. Secondary Outcome: Systolic BP
Description: Blood pressure was assessed using NCEP guidelines.
Time Frame: 6 months
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | A: EMPOWIR Diet and Placebo | B: EMPOWIR Diet Plus Metformin and Placebo Avandia | C: EMPOWIR Diet Plus Metformin and Avandia
Number analyzed (Participants) | 16 | 14 | 14
mmHg | 113.8 (2.9) | 107.2 (3.0) | 114.2 (4.7)
Statistical Analysis 1: Comparison: A: EMPOWIR Diet and Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.265, Paired t-test
Statistical Analysis 2: Comparison: B: EMPOWIR Diet Plus Metformin and Placebo Avandia; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.001, Paired t-test
Statistical Analysis 3: Comparison: C: EMPOWIR Diet Plus Metformin and Avandia; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.389, Paired t-test

6. Secondary Outcome: Diastolic BP
Description: Blood pressure was assessed using NCEP guidelines.
Time Frame: 6 months
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | A: EMPOWIR Diet and Placebo | B: EMPOWIR Diet Plus Metformin and Placebo Avandia | C: EMPOWIR Diet Plus Metformin and Avandia
Number analyzed (Participants) | 16 | 14 | 14
mmHg | 71.7 (2.3) | 72.7 (2.3) | 74.3 (3.8)
Statistical Analysis 1: Comparison: A: EMPOWIR Diet and Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.025, Paired t-test
Statistical Analysis 2: Comparison: B: EMPOWIR Diet Plus Metformin and Placebo Avandia; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.162, Paired t-test
Statistical Analysis 3: Comparison: C: EMPOWIR Diet Plus Metformin and Avandia; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.562, Paired t-test

7. Secondary Outcome: HDL
Description: HDL was measured using two reagents homogeneous systems with selective detergents to homogenize the lipoprotein of interest.
Time Frame: 6 months
Measure: Mean (Standard Error); unit: mg/dl
Arm/Group | A: EMPOWIR Diet and Placebo | B: EMPOWIR Diet Plus Metformin and Placebo Avandia | C: EMPOWIR Diet Plus Metformin and Avandia
Number analyzed (Participants) | 16 | 14 | 14
mg/dl | 56.5 (3.5) | 70.1 (5.8) | 68.3 (6.2)
Statistical Analysis 1: Comparison: A: EMPOWIR Diet and Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.016, Paired t-test
Statistical Analysis 2: Comparison: B: EMPOWIR Diet Plus Metformin and Placebo Avandia; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.03, Paired t-test
Statistical Analysis 3: Comparison: C: EMPOWIR Diet Plus Metformin and Avandia; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.150, Paired t-test

8. Secondary Outcome: Triglycerides
Description: Triglycerides were measured by enzymatic immunoassay on an AU400 chemistry auto-analyzer with commercially available enzymatic reagents.
Time Frame: 6 months
Measure: Mean (Standard Error); unit: mg/dl
Arm/Group | A: EMPOWIR Diet and Placebo | B: EMPOWIR Diet Plus Metformin and Placebo Avandia | C: EMPOWIR Diet Plus Metformin and Avandia
Number analyzed (Participants) | 16 | 14 | 14
mg/dl | 95.2 (10.7) | 103.1 (13.0) | 109.2 (18.3)
Statistical Analysis 1: Comparison: A: EMPOWIR Diet and Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.648, Paired t-test
Statistical Analysis 2: Comparison: B: EMPOWIR Diet Plus Metformin and Placebo Avandia; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.094, Paired t-test
Statistical Analysis 3: Comparison: C: EMPOWIR Diet Plus Metformin and Avandia; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.054, Paired t-test

9. Secondary Outcome: Adiponectin
Description: Total adiponectin was measured with a commercial ELISA kit (Millipore/Linco Research, St. Charles, MO) in the laboratory of Dr. Philipp Scherer.
Time Frame: 6 months
Measure: Mean (Standard Error); unit: ug/mL
Arm/Group | A: EMPOWIR Diet and Placebo | B: EMPOWIR Diet Plus Metformin and Placebo Avandia | C: EMPOWIR Diet Plus Metformin and Avandia
Number analyzed (Participants) | 16 | 14 | 14
ug/mL | 10.6 (1.2) | 10.9 (1.7) | 18.5 (1.5)
Statistical Analysis 1: Comparison: A: EMPOWIR Diet and Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.092, Paired t-test
Statistical Analysis 2: Comparison: B: EMPOWIR Diet Plus Metformin and Placebo Avandia; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.730, Paired t-test
Statistical Analysis 3: Comparison: C: EMPOWIR Diet Plus Metformin and Avandia; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Paired t-test

ADVERSE EVENTS:
Groups:
- A: EMPOWIR and Placebo: EMPOWIR dietary intervention food exchange program; 40-45% carbohydrates, 35-40% protein, and 20% fat AND 4 week dosage escalation of placebo metformin, 500 mg/day to a total dose of 2000mg/day; starting dose of placebo rosiglitazone 2mg/day added at weeks 3 and weeks 4 to a a total dose of 4 mg/day
- B: EMPOWIR Diet Plus Metformin and Placebo Avandia: EMPOWIR dietary intervention food exchange program; 40-45% carbohydrates, 35-40% protein, and 20% fat AND 4 week dosage escalation of metformin, 500 mg/day to a total dose of 2000mg/day; starting dose of rosiglitazone placebo 2mg/day added at weeks 3 and weeks 4 to a a total dose of 4 mg/day
- C: EMPOWIR Diet Plus Metformin and Avandia: EMPOWIR dietary intervention food exchange program; 40-45% carbohydrates, 35-40% protein, and 20% fat AND 4 week dosage escalation of metformin, 500 mg/day to a total dose of 2000mg/day; starting dose of rosiglitazone 2mg/day added at weeks 3 and weeks 4 to a a total dose of 4 mg/day
Arm/Group | A: EMPOWIR and Placebo | B: EMPOWIR Diet Plus Metformin and Placebo Avandia | C: EMPOWIR Diet Plus Metformin and Avandia
Serious Adverse Events (participants affected / at risk) | 1/16 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/16 | 0/15 | 0/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A: EMPOWIR and Placebo (N=16) | B: EMPOWIR Diet Plus Metformin and Placebo Avandia (N=15) | C: EMPOWIR Diet Plus Metformin and Avandia (N=15)
Worsening of Hypertension (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) — One patient with a prior history of hypertension was withdrawn due to elevated BP.

LIMITATIONS AND CAVEATS:
Widespread media coverage of cardiovascular risks of rosiglitazone led to an unanticipated high drop out rate of subjects just prior to their randomization; 22 of 68 eligible subjects did not undergo randomization due to concerns about the drug.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No